CLINICAL TRIAL: NCT06204302
Title: ARI Treatment Use and Outcomes in Non-metastatic Prostate Cancer (nmPC) Patients in the US
Brief Title: An Observational Study to Learn More About the Use of Androgen Receptor Inhibitors and How They Affect Men With Nonmetastatic Prostate Cancer in Routine Medical Care in the United States
Acronym: ARENA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22704
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Non-metastatic Prostate Cancer; Non-metastatic Castration-resistant Prostate Cancer
Keywords: nmPC; nmCRPC
MeSH Terms: interventions — darolutamide; enzalutamide; apalutamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Darolutamide: Participants with nmPC previously untreated with novel ARIs or abiraterone acetate and received Darolutamide as initial treatment.
  Interventions: Drug: Darolutamide (Nubeqa, BAY1841788)
- Enzalutamide: Participants with nmPC previously untreated with novel ARIs or abiraterone acetate and received Enzalutamide as initial treatment.
  Interventions: Drug: Enzalutamide
- Apalutamide: Participants with nmPC previously untreated with novel ARIs or abiraterone acetate and received Apalutamide as initial treatment.
  Interventions: Drug: Apalutamide

INTERVENTIONS:
Drug: Darolutamide (Nubeqa, BAY1841788) — Retrospective cohort analysis, using Komodo Research Database (KRD)
  Groups: Darolutamide
Drug: Enzalutamide — Retrospective cohort analysis, using Komodo Research Database (KRD)
  Groups: Enzalutamide
Drug: Apalutamide — Retrospective cohort analysis, using Komodo Research Database (KRD)
  Groups: Apalutamide

SUMMARY:
This is an observational study in which data will be collected and studied from men with non-metastatic prostate cancer (nmPC) who received their usual treatment with 'androgen receptor inhibitors' (ARIs) including darolutamide, enzalutamide, and apalutamide.

Prostate cancer is a common cancer in men that starts in the prostate gland, a male reproductive gland found below the bladder. Non-metastatic means that cancer has not yet spread to other parts of the body.

Darolutamide, enzalutamide, and apalutamide are already approved ARIs for nmPC in the United States (US). They work by blocking androgens (male sex hormones including testosterone) from attaching to proteins in cancer cells in the prostate. This helps to slow down the growth of the cancer cells. The participants will receive their treatments as prescribed by their doctors during routine medical care according to the approved product information.

Researchers want to know more about the use of ARIs and how they affect men with nmPC in the real world. Researchers will only include men who have not been treated with any new type of medication that blocks the action of male sex hormones.

The main purpose of this study is to collect and study information from men with nmPC about:

* the length of time they continued treatment with an ARI as prescribed by their doctors.
* the length of time from the start of the treatment with an ARI until the cancer spreads to other parts of the body.

Data will come from the participants' information stored in a database called Komodo Research Dataset (KRD) in the US.

The data collected will be from May 2019 to June 2023.

Researchers will only track data of eligible US men with nmPC and will follow them for a minimum of 6 months or until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Men diagnosed with prostate cancer (≥1 claim for prostate cancer).
* Treatment with apalutamide, darolutamide or enzalutamide initiated for the first time in the nmPC stage during the patient identification period.
* Age ≥ 18 years at index date
* At least 6 months of continuous eligibility in medical and pharmacy benefits prior to the index date
* At least 6-months of continuous eligibility only in pharmacy benefits after the index date unless patient died before 6 months.

Exclusion Criteria:

* Patients with multiple ARIs recorded at index date
* Use of an ARI agent or abiraterone acetate prior to the index date
* Other cancer diagnosis (except prostate and skin cancer) during the 6-month baseline period
* Evidence of metastatic disease any time before or 30 days after index date.
* No claim with a diagnosis for hormone sensitive malignancy status (Z19.1) during the study period

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men diagnosed with nmPC who were prescribed a novel ARI for the first time will be identified from Komodo Research Dataset (KRD) in the US.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Time to ARI discontinuation (days) for apalutamide, darolutamide, and enzalutamide | Retrospective analysis from index date 01 Aug 2019 up to 30 Jun 2023
Time to progression to metastatic prostate cancer (mPC) (days) for apalutamide, darolutamide, and enzalutamide | Retrospective analysis from index date 01 Aug 2019 up to 30 Jun 2023

SECONDARY OUTCOMES:
Descriptive summary of patient characteristics by cohort during baseline | Retrospective analysis from index date 01 May 2019 up to 31 Dec 2022
Descriptive summary of initiating prescribed daily dose of apalutamide, darolutamide, and enzalutamide | Retrospective analysis from index date 01 Aug 2019 up to 30 Jun2023
Descriptive summary of initiating prescribed daily dose intensity of apalutamide, darolutamide, and enzalutamide | Retrospective analysis from index date 01 Aug 2019 up to 30 Jun2023
Initiating dose changes (increase/decrease) of apalutamide, darolutamide, and enzalutamide (yes/no) | Retrospective analysis from index date 01 Aug 2019 up to 30 Jun2023
Switching between apalutamide, darolutamide, and enzalutamide (yes/no) | Retrospective analysis from index date 01 Aug 2019 up to 30 Jun2023
Proportion of days covered (PDC) | Retrospective analysis from index date 01 Aug 2019 up to 30 Jun2023
  PDC is calculated by dividing the total non-overlapping days of supply by the length of a fixed time interval (6, 12, 18, 24 months) and by the patient specific treatment duration.

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer, Whippany, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.